CLINICAL TRIAL: NCT00788320
Title: Antimicrobial Peptide LL-37 (Cathelicidin) Production in Active Tuberculosis Disease: Role of Vitamin D Supplementation
Brief Title: Vitamin D in Active Tuberculosis (TB) Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vin Tangpricha, Associate Professor, Atlanta VA Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vitamin D in TB
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; vitamin D; immune system
MeSH Terms: conditions — Tuberculosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo three times a week for 8 weeks
  Interventions: Drug: Placebo
- Cholecalciferol (Experimental): Vitamin D3 50,000 IU three times a week for 8 weeks
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 50,000 IU three times a week for 8 weeks
  Arms: Cholecalciferol
Drug: Placebo — Placebo three times a week for 8 weeks
  Arms: Placebo

SUMMARY:
Tuberculosis is a disease caused by a bacterium (a germ) that can cause illness in any organ of the body, but most frequently causes disease of the lungs. TB is short for tuberculosis. Treating TB requires several months (usually 6 months) of treatment, with the first 2 months being intensive treatment with usually four medicines. Treatment is needed to keep the infection from getting worse and to prevent death from TB.

Vitamin D is a hormone present in the human body to manage levels of some essential electrolytes such as calcium and phosphate. Vitamin D is important for bone formation and prevention of bone breakdown (osteoporosis) as the investigators age. There is also new evidence that links vitamin D to function of our immune system as well. Even though our bodies can make vitamin D and can also obtain vitamin D from our diet, most adults, especially patients with tuberculosis have low vitamin D levels (are vitamin D deficient) that need to be corrected. Full correction of low vitamin D levels requires 6 weeks or more of weekly vitamin D supplements. There are several benefits to correcting vitamin D deficiency (better bone health, better balance of calcium and phosphate), but it is not known whether correcting vitamin D deficiency will lead to a better immune response to tuberculosis. Preliminary data does suggest that vitamin D increases the levels of an antimicrobial molecule (cathelicidin LL-37) in the body, possibly leading to better immunity against tuberculosis. The primary objective of this pilot study is to assess the relationship of vitamin D levels in patients with active pulmonary tuberculosis to levels of LL-37 cathelicidin in sputum and whole blood. The results of this study are needed in preparation for larger studies that will evaluate the role of vitamin D supplementation as adjunctive therapy to standard medical treatment for tuberculosis.

DETAILED DESCRIPTION:
1.0 Introduction and Background

Tuberculosis remains an enormous public health problem and a major cause of morbidity and mortality throughout the world. The WHO estimates that 8.8 million new cases of tuberculosis occurred worldwide in 2005, along with 1.6 million TB related deaths. New challenges in TB control include the HIV epidemic, as well as the emergence of multidrug resistant (MDR) and extremely drug resistant (XDR) strains of tuberculosis which are associated with high morbidity and mortality. While cure rates for drug susceptible TB can reach the >90% range given the appropriate infrastructure to diagnose and treat patients, cure rates for MDR-TB are much lower and, at best, approach 60% according to the latest estimates by WHO. In many parts of the world, second line drugs to treat MDR-TB are not available. Not only is there an urgent need for novel TB treatment regimens, but adjunctive therapeutic modalities need to be explored with the goal of maximizing clinical response for both patients with drug susceptible and drug resistant disease.

The use of vitamin D as primary or adjunctive TB therapy has a long history. Therapeutic doses of oral vitamin D supplementation for TB treatment were first pioneered in the 1950's by Jacques Charpy, who noted excellent results in cutaneous TB disease. Subsequently, vitamin D has been used as both primary and adjunctive therapy in pulmonary tuberculosis, but this practice fell out of favor as effective antimycobacterial chemotherapy became widely available in the latter half of the twentieth century.

More recently, however, there has been a resurgence of interest in vitamin D as an effective adjunctive therapy in tuberculosis. Recent reports indicate that vitamin D may have a pronounced immunomodulatory role in the pathogenesis of tuberculosis within the human host. It is well known that areas of granulomatous inflammation in TB are sites of increased vitamin D production stemming from activated macrophages and Th1 lymphocytes within the granuloma Recently, the immunomodulatory function of increased vitamin D levels at sites of TB involvement has been demonstrated, in that 1,25(OH)2D, the active metabolite form of vitamin D, has been found to induce antimycobacterial activity in vitro in both monocytes and macrophages.

One proposed pathway for this observed immunomodulatory effect of vitamin D in TB infection involves the toll-like receptor (TLR) signaling pathways of the innate immune system. Liu et al demonstrated that macrophage TLR binding of M. tuberculosis antigen upregulates the expression of cellular 1 hydroxylase, resulting in higher levels of active 1, 25(OH)2D. It was also shown that 1, 25(OH)2D in turn binds the nuclear vitamin D receptor (VDR), which activates a downstream signaling cascade resulting in the upregulation of several aspects of the innate immune response, including the induction of a newly described anti-microbial peptide LL-37, a cathelicidin. Cathelicidins, in addition to their broad spectrum antimicrobial activity, also possess chemotactic properties for neutrophils, monocytes and T cells, among other functions within the immune system.

While this mechanism of action for vitamin D was demonstrated in vitro, little clinical work has been done to validate this piece of knowledge in clinical practice and in the care of TB patients. As proxy for in vivo studies, subsequent experiments by Liu et al evaluated induction of cathelicidin by TLR activation of macrophages in sera from African American and Caucasian subjects. These experiments demonstrated failure to induce detectable levels of cathelicidin mRNA in samples from African American patients, who are known to be significantly more vitamin D deficient than Caucasians due to difference in vitamin D production in the skin. The difference in cathelicidin mRNA levels was corrected upon supplementation of deficient sera to therapeutic levels of 25(OH)D3 prior to TLR stimulation.

Given the preliminary results of these in vitro studies, we propose a clinical pilot investigation of the relationship between vitamin D levels and cathelicidin production in TB patients. It is well known that the majority of TB patients are deficient in vitamin D, but it is unknown whether the deficiency has functional consequences for treatment response and relapse rates. While recent in vitro data suggests that vitamin D supplementation of recent TB contacts does improve their immune response to Mycobacterium tuberculosis as measured in whole blood assays, clinical trials of vitamin D supplementation in latent or active TB disease have not been undertaken. In preparation for larger trials that would be needed to address this clinical question, we propose that the clinical relationship between physiologic levels of vitamin D supplementation and effect on cathelicidin production within the host needs to be studied, given recent suggestions from in vitro studies that ability to generate adequate cathelicidin levels may have an impact on quality and effectiveness of host immune defense against M. tuberculosis.

2.0 Objectives

2.1 Overall Objective

The primary objective of this pilot study is to assess the relationship of 25-hydroxy vitamin D levels in patients with active pulmonary tuberculosis to levels of LL-37/cathelicidin in sputum, saliva, and whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must be patients with newly diagnosed laboratory confirmed pulmonary tuberculosis (i.e., no previous history of treatment for TB for more than 30 days). Those enrolled should not have received more than 1 week of antituberculosis therapy prior to enrollment.
* Study subjects must agree to participate in the study and provide written informed consent
* Histology: not applicable
* Sites: Emory University affiliated hospitals (including Emory University Hospital, Emory Crawford Long Hospital, Grady Memorial Hospital), and metropolitan Atlanta health departments including the Fulton County Department of Health and Wellness and the DeKalb County Board of Health as well as additional health departments in the Metropolitan Atlanta area.
* Stage of Disease: pulmonary tuberculosis patients who have completed less than 1 week of TB therapy
* Age: Study subjects must be > 18 years old
* Performance Status: study subjects will be patients with newly diagnosed laboratory confirmed pulmonary TB who have completed < 1 week of anti-TB therapy and who are able to provide written informed consent
* Informed consent requirements: All study subjects must agree to participate in the study and provide written informed consent, which will be written in English. An additional consent form will be provided to subjects who agree to long term storage of their blood, saliva, and sputum samples for future use by the investigators of this study. For subjects who do not speak English, a short consent form will be used to obtain informed consent, which will be available in the the 10 most commonly encountered languages in the greater Atlanta area after English. The short form will be used in conjunction with an interpreter who will assist in translating and discussing the content of the long form prior to the subjects' signing of the short form.

Exclusion Criteria:

* Age < 18years
* Prior anti-microbial drug treatment of tuberculosis for longer than 1 week
* Prior other diseases: patients with prior disorders potentially affecting vitamin D levels and metabolism of calcium and phosphate will be excluded. Pregnant or lactating women are ineligible for this study. We plan to exclude patients with any known disorders of the endocrine system affecting vitamin D metabolism, including: hyperparathyroidism, known history of nephrolithiasis, any documented malignancies, and advanced renal disease. Patients with prior disorders that may potentially affect cathelicidin levels will be excluded as well. These diseases include atopic dermatitis (eczema) and hematologic malignancies (leukemia, lymphoma, among others)
* Infection: not applicable
* Hematologic, renal and hepatic, and other values that preclude entry into the study: serum creatinine of >1.5 mg/dL to assist with exclusion of patients with renal disease. Patients with baseline calcium level >10.5 mg/dL will be excluded to assist with exclusion of pre-existing disorders of vitamin D and calcium metabolism (see Section C above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
LL-37 level | 8 weeks

SECONDARY OUTCOMES:
Sputum Conversion | 8 weeks
25-hydroxyvitamin D and serum calcium | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States